CLINICAL TRIAL: NCT03074461
Title: Transverse Coloplasty vs. Side-to-end Anastomosis Following Low Anterior Resection (LAR): CSAR Trial
Acronym: CSAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Markus Rentsch, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-129
Record Dates: First submitted 2017-02-26; First posted 2017-03-08 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Rectal Cancer; Rectal Neoplasms; Rectal Tumors; Fecal Incontinence
Keywords: Rectal Cancer; Low Anterior Resection; Coloplasty Pouch; Side-to-end Anastomosis; Continence; Quality of Life
MeSH Terms: conditions — Rectal Neoplasms; Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized in two parallel study arms regarding their neorectal reconstruction in low anterior resection, the experimental arm using the side-to-end anastomosis and the control group using the transverse coloplasty technique.
Masking Description: There is no masking in the CSAR Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side-to-End (Experimental): Side-to-End Anastomosis as neorectal reconstruction technique in low anterior resection (LAR)
  Interventions: Procedure: Side-to-End Anastomosis
- Transverse Coloplasty (Active Comparator): Transverse Coloplasty pouch as neorectal reconstruction technique in low anterior resection (LAR)
  Interventions: Procedure: Transverse Coloplasty

INTERVENTIONS:
Procedure: Side-to-End Anastomosis — During the scheduled low anterior resection (LAR) in patients with distal rectal cancer and anticipated anastomosis in the mid or distal rectal third, the reconstruction phase of the LAR consists of the implementation of a side-to-end colorectal anastomosis.
  Arms: Side-to-End
Procedure: Transverse Coloplasty — During the scheduled low anterior resection (LAR) in patients with distal rectal cancer and anticipated anastomosis in the mid or distal rectal third, the reconstruction phase of the LAR consists of the implementation of a transverse coloplasty pouch. For this purpose an end-to-end colorectal anastomosis is initially performed, followed by a longitudinal incision of approx. 8-10 cm length proximal of the anastomosis and a subsequent transverse suture in terms of the coloplasty technique.
  Other Names: Coloplasty Pouch, Transverse Coloplasty Pouch
  Arms: Transverse Coloplasty

SUMMARY:
CSAR Trial's aim is to determine whether the transverse coloplasty pouch or the side-to-end anastomosis as rectal reservoir reconstruction offers the best functional results.

DETAILED DESCRIPTION:
This study directly compares two neorectal reservoir-techniques, the transverse coloplasty and the side-to-end anastomosis, in low anterior resection in distal rectal cancer for the first time. Its focus is on the functional results. Besides stool frequency, the quality of life, safety of the procedures and the usage of stool modulating drugs is monitored in an 12 months-follow up regime.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled low anterior resection in patients with distal rectal carcinoma and planned anastomosis in mid/distal third of rectum
* Local curative approach
* Normal continence preoperatively
* Non-IBD-associated carcinoma
* Possible sphincter salvage
* Signed informed consent

Exclusion Criteria:

* Non-curative approaches
* Emergency surgery in cases of tumor perforation, abscess, sepsis
* Proximal rectal carcinoma (> 12 cm from anocutaneous line)
* Lack of informed consent
* Age <18 years
* Inclusion in other trials with interference of endpoints
* Life expectancy less than 24 months (as estimated by the treating physicians)
* Pregnancy
* Immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Stool frequency | time = 6 months postoperative
  Between group differences in stool frequency at t = 6 months postoperative

SECONDARY OUTCOMES:
Postoperative complications | through study completion (an average of 12 months postoperative)
  * Septic intraabdominal complications related to anastomosis (anastomotic insufficiencies, suture insufficiencies, abscesses);
  * Wound infection
Quality of Life | baseline, postoperative (2-3 months, 6 months, 12 months)
  Quality of Life with focus on colorectally specialized questionnaires
Antimotility drug usage | baseline, postoperative (2-3 months, 6 months, 12 months)
  Usage of antimotility drugs (e.g. loperamide) evaluated by standardized questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Markus Rentsch, MD, Principal Investigator — Department of General, Visceral, and Transplantation Surgery
Locations (3):
- Germany (3):
  - Maria-Theresia-Klinik, München, Bavaria
  - Krankenhaus Barmherzige Brüder München, München, Bavaria
  - Klinikum der Universität München, München, Bavaria

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to third parties beyond the study team.